CLINICAL TRIAL: NCT02803502
Title: Does the Thrombin Generation Test Performed During the Pharmacokinetic Profile of the Substitutive Factor VIII Bring Benefits to the Personalized Treatment of Pediatric Patients and Adult Hemophilia A Patients Under Prophylaxis ?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Dr Anne Demulder, Head of clinic, Brugmann University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHUB-PK TGT
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Hemophilia
Keywords: thrombin generation test; factor VIII; hemophilia
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hemophilia (Experimental): Patients with severe hemophilia (or moderate hemophilia if presence of hemorrhages) under prophylaxy and subjected to a pharmacokinetic profile of factor VIII
  Interventions: Device: Chronometric method; Device: Chromogenic method; Device: Thrombin generation test (TGT)

INTERVENTIONS:
Device: Chronometric method — Chronometric method of FVIII dosage on STA-R PLC automate (reactive Cephascreen STAGO, Unicalibrateur STAGO, plasma deficient Cryopep, Controls STAGO)
Device: Chromogenic method — Chromogenic FVIII assay method ( "BIOPHEN FVIII: C" and "BIOPHEN Factor IX" of the firm Hyphen BioMed)
Device: Thrombin generation test (TGT) — Briefly: the measurement of thrombin generation is performed by the technique of calibrated and automated Thrombinography (CAT) developed by Hemker HC. This technique allows the simultaneous analysis of multiple samples using a fluorometer (Fluoroscan Ascent, ThermoLabsystems OY, Helsinki, Finland) and a Thrombinoscope® software that converts the fluorescence intensity obtained by concentration of active thrombin. The reagent "PPP-reagent Low" respectively containing 1pm FT and 4μM phospholipid (PL) as a final concentration will be used.

SUMMARY:
In the context of hemophilia, it is well know that the level of factor VIII alone does not reflect the clinical phenotype of the patients in an accurate way. At equal factor VIII levels, certain patients will bleed more than others.

The thrombin generation test (TGT) is a test that seems to provide a better prediction of the overall hemostatic status of an individual patient. In a previous study, the investigators have established normal reference values of the thrombin generation curve in children aged 6 months to 16 years and adults. The goal was to evaluate the use of this test in different clinical contexts and in severe hemophilia patients in particular. A pilot study showed that the patients having a thrombin generation <150 had a severe phenotype, whether those who received an appropriate prophylaxy had a thrombin generation superior to 150.

Moreover, the investigators now have access to a software tool that allows them to individually determine the pharmacokinetic profile of the factor VIII injected to each patient. The factor VIII concentration is measured at injection and 30 minutes, 1 hour, 2 hours and 24 hours afterwards. The introduction of these concentrations in the software allows to obtain the half-life of factor for a given patient, the maximum peak, and the minimum factor level (though level). The injected dosis might be sufficient (disappearance of substantial diminution of the bleedings) or unsufficient (persisting bleeding) for a given patient.

This study aims:

* to measure the pharmacokinetic profile of factor VIII by two different methods, the time-based method and the chromogenic method
* to correlate the results with the TGT results obtained at the same time points and determine which method gives the best correlation
* to link the clinical symptomatology (improved symptomatology or not) with the TGT results
* to determine which minimal TGT result is linked to a minimal bleeding rate
* to adapt the prophylactic dosis of the patient in a personalized way.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe or moderate hemophilia, on prophylaxis, and suffering from bleedings.

Exclusion Criteria:

* Patients with difficult venous access
* Patients who have had surgery or trauma in the month before, patients with acute disease (infection, inflammation)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Factor VIII blood concentration - chronometric method | baseline: at factor VIII injection
  Chronometric method of FVIII dosage on STA-R PLC automate (reactive Cephascreen STAGO, Unicalibrateur STAGO, plasma deficient Cryopep, Controls STAGO)
Factor VIII blood concentration - chronometric method | 30 minutes after factor VIII injection
  Chronometric method of FVIII dosage on STA-R PLC automate (reactive Cephascreen STAGO, Unicalibrateur STAGO, plasma deficient Cryopep, Controls STAGO)
Factor VIII blood concentration - chronometric method | 60 minutes after factor VIII injection
  Chronometric method of FVIII dosage on STA-R PLC automate (reactive Cephascreen STAGO, Unicalibrateur STAGO, plasma deficient Cryopep, Controls STAGO)
Factor VIII blood concentration - chronometric method | 120 minutes after factor VIII injection
  Chronometric method of FVIII dosage on STA-R PLC automate (reactive Cephascreen STAGO, Unicalibrateur STAGO, plasma deficient Cryopep, Controls STAGO)
Factor VIII blood concentration - chronometric method | 24h after factor VIII injection
  Chronometric method of FVIII dosage on STA-R PLC automate (reactive Cephascreen STAGO, Unicalibrateur STAGO, plasma deficient Cryopep, Controls STAGO)
Factor VIII blood concentration - Chromogenic method | baseline: at factor VIII injection
  Chromogenic FVIII assay method ( "BIOPHEN FVIII: C" and "BIOPHEN Factor IX" of the firm Hyphen BioMed)
Factor VIII blood concentration - Chromogenic method | 30 minutes after factor VIII injection
  Chromogenic FVIII assay method ( "BIOPHEN FVIII: C" and "BIOPHEN Factor IX" of the firm Hyphen BioMed)
Factor VIII blood concentration - Chromogenic method | 60 minutes after factor VIII injection
  Chromogenic FVIII assay method ( "BIOPHEN FVIII: C" and "BIOPHEN Factor IX" of the firm Hyphen BioMed)
Factor VIII blood concentration - Chromogenic method | 120 minutes after factor VIII injection
  Chromogenic FVIII assay method ( "BIOPHEN FVIII: C" and "BIOPHEN Factor IX" of the firm Hyphen BioMed)
Factor VIII blood concentration - Chromogenic method | 24h after factor VIII injection
  Chromogenic FVIII assay method ( "BIOPHEN FVIII: C" and "BIOPHEN Factor IX" of the firm Hyphen BioMed)
total thrombin generation | baseline: at factor VIII injection
  the measurement of thrombin generation is performed by the technique of calibrated and automated Thrombinography (CAT) developed by Hemker HC. This technique allows the simultaneous analysis of multiple samples using a fluorometer (Fluoroscan Ascent, ThermoLabsystems OY, Helsinki, Finland) and a Thrombinoscope® software that converts the fluorescence intensity obtained by concentration of active thrombin.
total thrombin generation | 30 minutes after factor VIII injection
  the measurement of thrombin generation is performed by the technique of calibrated and automated Thrombinography (CAT) developed by Hemker HC. This technique allows the simultaneous analysis of multiple samples using a fluorometer (Fluoroscan Ascent, ThermoLabsystems OY, Helsinki, Finland) and a Thrombinoscope® software that converts the fluorescence intensity obtained by concentration of active thrombin.
total thrombin generation | 60 minutes after factor VIII injection
  the measurement of thrombin generation is performed by the technique of calibrated and automated Thrombinography (CAT) developed by Hemker HC. This technique allows the simultaneous analysis of multiple samples using a fluorometer (Fluoroscan Ascent, ThermoLabsystems OY, Helsinki, Finland) and a Thrombinoscope® software that converts the fluorescence intensity obtained by concentration of active thrombin.
total thrombin generation | 120 minutes after factor VIII injection
  the measurement of thrombin generation is performed by the technique of calibrated and automated Thrombinography (CAT) developed by Hemker HC. This technique allows the simultaneous analysis of multiple samples using a fluorometer (Fluoroscan Ascent, ThermoLabsystems OY, Helsinki, Finland) and a Thrombinoscope® software that converts the fluorescence intensity obtained by concentration of active thrombin.
total thrombin generation | 24h after factor VIII injection
  the measurement of thrombin generation is performed by the technique of calibrated and automated Thrombinography (CAT) developed by Hemker HC. This technique allows the simultaneous analysis of multiple samples using a fluorometer (Fluoroscan Ascent, ThermoLabsystems OY, Helsinki, Finland) and a Thrombinoscope® software that converts the fluorescence intensity obtained by concentration of active thrombin.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Demulder, MD, Principal Investigator — CHU Brugmann
Locations (5):
- Belgium (5):
  - CHU Brugmann, Brussels
  - HUDERF, Brussels
  - Centre Hospitalier Régional de la Citadelle de Liège, Liège
  - CHC de Liège, Liège
  - CHU Liège Sart Tilman, Liège

REFERENCES:
- [Background] Hemker HC, Giesen P, AlDieri R, Regnault V, de Smed E, Wagenvoord R, Lecompte T, Beguin S. The calibrated automated thrombogram (CAT): a universal routine test for hyper- and hypocoagulability. Pathophysiol Haemost Thromb. 2002 Sep-Dec;32(5-6):249-53. doi: 10.1159/000073575. PMID 13679651
- [Background] Filippin L, Debaugnies F, Noubouossie D, Le PQ, Ferster A, Demulder A. [Thrombin generation test: establishment of reference values according to age and tissue factor concentration is essential before implementation into the laboratory]. Rev Med Brux. 2011 Mar-Apr;32(2):69-73. French. PMID 21688590
- [Background] van den Berg HM, De Groot PH, Fischer K. Phenotypic heterogeneity in severe hemophilia. J Thromb Haemost. 2007 Jul;5 Suppl 1:151-6. doi: 10.1111/j.1538-7836.2007.02503.x. PMID 17635721